CLINICAL TRIAL: NCT05258201
Title: Effect of Muscle Energy Technique Versus Strain-Counterstrain on Upper Trapezius Myofascial Active Trigger Points. A Randomized Control Trial
Brief Title: Effect of Muscle Energy Technique Versus Strain-counterstrain on Upper Trapezius Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-FSD-00268
Record Dates: First submitted 2022-02-20; First posted 2022-02-28 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Trigger Point Pain, Myofascial
Keywords: Muscle Energy Technique; Myofascial; Trigger Point; Upper Trapezius; Strain-counterstrain
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Our study will be single-blinded, outcome assessor-blinded. The assessor will be blinded to avoid being biased during the outcome assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle Energy Technique (Experimental): Muscle energy Technique will be applied on the subjects, when they will be lying supine and on the effect side therapist will stabilize shoulder by one hand, while the ear / mastoid area of the affected side will be hold by opposite hand. The head and neck will be bend to contralateral side, then bends on the same side. Subject will raise his shoulder with the shoulder fixed to the ear with less effort than the maximum. Isometric contraction will be maintain for 7-10 seconds. This position will be held for 30 seconds and repeat three to five times per on treatment session
  Interventions: Other: Muscle Energy Technique
- Strain-counterstrain (Experimental): Strain And Counter Strain will be applied on subject in normal position and will be produced by placing the muscle in a short / relaxed position, the point where the pain will reduce of at least 70% will be produce will easily define. The patient will be in a supine position while the doctor will place the labial arm in flexion, abduction and external rotation to reduce the reported Trp pain. Once the position is easy to find, the pressure will be apply to the Trp and will be hold for 20-30 seconds and repeat this process for up to five times
  Interventions: Other: Strain-counterstrain

INTERVENTIONS:
Other: Strain-counterstrain — Strain-counterstrain is also used for manual Trigger Point processing. This involves identifying active TRP and then applying pressure until a ridiculous reaction occurs. The area is then positioned to reduce tension in the injured muscle and later reduce tripod pain. When the pain subsides, the tissues that are most stressed feel relaxed and there is a local decrease in the ground
  Arms: Strain-counterstrain
Other: Muscle Energy Technique — Muscle Energy Technique is a common way to achieve muscle tension release (stop) before stretching other's adductor muscles
  Arms: Muscle Energy Technique

SUMMARY:
Aim of the study To determine the comparative effects of muscle energy technique and strain counter strain in upper trapezius trigger point.

DETAILED DESCRIPTION:
A Randomized Controlled trial will be conducted after approval of synopsis. To enroll patients Purposive sampling technique will be used. Patients will be selected according to the pre-defined inclusion and exclusion criteria. The enrolled patients will be allocated into two groups, group A and group B. On Group A muscle energy technique will be applied for 30 seconds and repeat 3 to 5 times per on treatment session and Group B will be treated with strain counter strain for 20-30 seconds and repeat this process for up to five times. Assessment will be done at baseline, 2nd week, 4th week and 6th week of treatment. Follow up will be assessed 15 days after completion of treatment protocol. The patients' outcome will be measured by Visual Analog Scale for pain intensity and Neck Disability Index . Informed consent will be taken from each patient. Statistical Package of Social Sciences software, version 20 will be used for the analysis of data.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are 18 to 34 years old
2. In upper trapezius From 2 weeks Had mechanical neck pain and was diagnosed with active myofacial Trigger points
3. Subjects have to exhibit a tendor point in the upper trapezius muscle either on the left or right side
4. Local pain is greater than 3/10 on Visual Analog scale

Exclusion Criteria:

1. Patient with cervical radiculopathy
2. Patients with Fibromyalgia syndrome
3. Patients who had cervical spine surgery
4. Patient with myelopathy
5. Patients who had myofacial pain therapy

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 12th Week
  A Visual Analogue Scale is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms.
Neck Disability Index | 12th Week
  The Neck Disability Index is a 10-item questionnaire that measures a patient's self-reported neck pain related disability. A higher Neck Disability Index score means the greater a patient's perceived disability due to neck pain
Goniometer | 12th Week
  Goniometer has been the most widely used tool for measuring joint range of motion. To ensure reliable measurement, standardized, specific positions and landmarks are used to measure Cervical lateral flexion range of motion.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No